CLINICAL TRIAL: NCT05734092
Title: Investigating the Effectiveness of Low-Level Laser in Reducing Root Resorption of the Upper Incisors During Intrusion Movement Using Mini-Implants in Adult Patients With Deep Overbite: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Root Resorption During the Correction of Deep Bite With the Help of Laser Irradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-02-2023
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Deep Overbite
Keywords: Low-level laser; Deep bite; Mini-implants; Root resorption
MeSH Terms: conditions — Overbite; Root Resorption | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The strength of the nickel-titanium coil will be adjusted every 4 weeks to the required strength of 40 g on each end until reaching normal coverage
  Interventions: Device: Traditional orthodontic treatment
- Low-Level Laser Therapy group (Experimental): In the experimental group (LLLT), where a (Ga-Al-As) diode laser, will be used with 808 nm wavelength in continuous mode, 250 milli-Watt power output, 4 Joules/point energy density, 16 s per point. In addition to adjusting the force gauge every 4 weeks until the end of the intrusion stage and reaching normal coverage
  Interventions: Device: Low-Level Laser

INTERVENTIONS:
Device: Traditional orthodontic treatment — As for patients in the control group, the strength of the nickel-titanium coil will be adjusted every 4 weeks to the required strength of 40 g on each end until reaching normal coverage.
  Arms: Control group
Device: Low-Level Laser — The laser will be applied to the root of each of the upper incisors in 8 points (4 points from the labial and 4 points from the palatine), and the head of the device will be placed from the labial side of the root in the center of each of the apical and middle thirds and the mesial and distal of the cervical third in contact with Oral mucosa perpendicular to the root axis, with the application of the laser beam for (16) seconds at one point, and the laser will be re-applied in the same way from the palatal side of the root. So that it was the total application time is (128) seconds for one tooth.
  The laser will be applied on the day the upper incisor intrusion started (T1), then on days (3, 7, and 14) of the first month, and starting from the second month, the laser will be applied every (15) day, in addition to adjusting the force gauge every 4 weeks until the end of intrusion stage (T2) and reaching normal coverage.
  Arms: Low-Level Laser Therapy group

SUMMARY:
This study aims to investigate the effectiveness of low-level laser in reducing the resorption of the roots of the upper incisors. Participants will be recruited from patients who will attend the Department of Orthodontics and Dentofacial Orthopaedics at Damascus University. The study sample will consist of 30 patients with a deep bite who will be randomly distributed equally into two groups, 15 patients in each group, average age: 22.37±3.38 years. Mini-implants will apply between the roots of the maxillary central and lateral incisor at both sides with a loading force of 40 g on each end by using a nickel-titanium spring extending from the head of the mini-implants to a wire welded to it with two hooks. A low-level laser (Ga-Al-As) will be used with 808 nm wavelength in continuous mode, 250 milli-Watt power output, 4 Joules/point energy density, 16 s per point in the experimental group. It will be applied on the day of intrusion, then on days 3,7, and 14 of the first month, and then every 15 days starting from the second month until the end of the intrusion. In addition to adjusting the force gauge every 4 weeks until the end of the intrusion stage and reaching normal coverage will be activated every 4 weeks in both groups until normal overbite was reached.

DETAILED DESCRIPTION:
Several studies have indicated the effectiveness of the LLLT in accelerating orthodontic movement, but studies that have evaluated the role of this laser in reducing the risk of OIIRR have been limited. Moreover, the effects of laser in reducing root resorption have been studied with different types of orthodontic movements such as en masse anterior retraction, canine retraction, and tilting of the premolars before extraction, but they have not been studied with the intrusion movement

ELIGIBILITY:
Inclusion Criteria:

1. overbite > 4 mm
2. Class I or II molar and canine relationship malocclusion
3. maxillary anterior crowding < 2 mm
4. maxillary incisors positioned below the functional occlusal plane
5. incisor display of 2-3 mm or more at rest
6. the facial growth pattern is normal or horizontal.

Exclusion Criteria:

1. the maxillary incisors had a history of any trauma or endodontic treatment
2. increased inclination of the maxillary incisors towards the labial
3. the subject had any systemic disease
4. the patient exhibited poor oral hygiene

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change in root volume | T1: One day before the beginning of the incisor intrusion procedure, T2: One day following the end of the incisor intrusion procedure which is expected to happen within 4 to five months.
  The root volume will be measured using cone-beam computed tomography (CBCT) images.
  One CBCT image will be taken before starting the incisor intrusion Another image will be taken after the end of intrusion (which is expected to happen within 4 to 5 months) Each root's volume will be calculated using specific software (Mimics 21.0, Materialise NV Technologielaan, Leuven).
  This calculation will be performed for the upper incisors (central and lateral incisors).
Change in root length | T1: One day before the beginning of the incisor intrusion procedure, T2: One day following the end of the incisor intrusion procedure which is expected to happen within 4 to five months.
  The root volume will be measured using cone-beam computed tomography (CBCT) images (employing the sagittal view).
  One CBCT image will be taken before starting the incisor intrusion Another image will be taken after the end of intrusion (which is expected to happen within 4 to 5 months) Each root's length will be calculated using the 3D viewing software. This calculation will be performed for each tooth in the upper anterior region; i.e., upper central and lateral incisors.

CONTACTS AND LOCATIONS:
Overall Officials: Amer Ramez Nasser, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Kinda Sultan, DDS MSc PhD, Study Director — Department of orthodontics, Damascus University, Syria; Mohammad Y. Hajeer, DDS MSc PhD, Study Director — Department of orthodontics, Damascus University, Syria; Omar Hamadah, DDS MSc PhD, Study Director — Department of oral medicine, Damascus University, Syria
Locations (1):
- Mohammad Y. Hajeer, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng D, Chan AK, Papadopoulou AK, Dalci O, Petocz P, Darendeliler MA. The effect of low-level laser therapy on orthodontically induced root resorption: a pilot double blind randomized controlled trial. Eur J Orthod. 2018 May 25;40(3):317-325. doi: 10.1093/ejo/cjx065. PMID 29016741
- [Background] Jaber ST, Al-Sabbagh R, Hajeer MY. Evaluation of the efficacy of laser-assisted flapless corticotomy in accelerating canine retraction: a split-mouth randomized controlled clinical trial. Oral Maxillofac Surg. 2022 Mar;26(1):81-89. doi: 10.1007/s10006-021-00963-x. Epub 2021 Apr 20. PMID 33876339
- [Background] Ang Khaw CM, Dalci O, Foley M, Petocz P, Darendeliler MA, Papadopoulou AK. Physical properties of root cementum: Part 27. Effect of low-level laser therapy on the repair of orthodontically induced inflammatory root resorption: A double-blind, split-mouth, randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2018 Sep;154(3):326-336. doi: 10.1016/j.ajodo.2018.04.022. PMID 30173835
- [Background] Aras I, Tuncer AV. Comparison of anterior and posterior mini-implant-assisted maxillary incisor intrusion: Root resorption and treatment efficiency. Angle Orthod. 2016 Sep;86(5):746-52. doi: 10.2319/085015-571.1. Epub 2016 Jan 7. PMID 26741306
- [Background] Altan AB, Bicakci AA, Mutaf HI, Ozkut M, Inan VS. The effects of low-level laser therapy on orthodontically induced root resorption. Lasers Med Sci. 2015 Nov;30(8):2067-76. doi: 10.1007/s10103-015-1717-6. Epub 2015 Jan 30. PMID 25633918